CLINICAL TRIAL: NCT04343040
Title: Perioperative Evaluation of Glucose Profile Using Continuous Glucose Monitoring System in Glucose Intolerant Patients Submitted to Bariatric Surgery and Receiving Pre-operative Carbohydrate Loading in Comparison With Standard 6h Fasting - A Single Center, Open-label, Randomized Pilot Study
Brief Title: Perioperative Evaluation of Glucose Profile Using Continuous Glucose Monitoring System in Glucose Intolerant Patients
Acronym: PERISURG-CGM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017_34; 2017-A03320-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-04-06; First posted 2020-04-13 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Hyperglycaemia (Diabetic); Bariatric Surgery Candidate
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perioperative glucose intake (Experimental): glucose intolerant patients with perioperative glucose (carbohydrate supplement (Preload™) intake before Gastric By-Pass or Sleeve Gastrectomy.
  Interventions: Dietary Supplement: carbohydrate supplement (Preload™)
- 6 hours of preoperative fasting (Sham Comparator): glucose intolerant patients receiving 6 hours of preoperative fasting before Gastric By-Pass or Sleeve Gastrectomy.
  Interventions: Procedure: 6 hours of preoperative fasting

INTERVENTIONS:
Dietary Supplement: carbohydrate supplement (Preload™) — carbohydrate supplement (Preload™) will be administered 4-hours prior to bariatric surgery (experimental treatment) Preload™ is a neutral-tasting carbohydrate loading drink mix specifically designed for use before elective surgery. Preload is presented in 50g pre-measured sachets which when added to water (400ml) produces a solution with low osmolality.
  Arms: perioperative glucose intake
Procedure: 6 hours of preoperative fasting — Standard of care. In this group, patients continue the standard of care treatment before surgery with fasting recommended 6 hours before surgery.
  Arms: 6 hours of preoperative fasting

SUMMARY:
The recent use of a pre-operative carbohydrate loading compared to fasting has been shown to improve the early recovery after surgical procedures by reducing the profound stress response following surgery and allowing a better postoperative blood glucose regulation by lowering insulin resistance. The responsible mechanisms of T2D remission after bariatric surgery are not completely understood and guidelines for the early management of T2D and GI following bariatric surgery are lacking, resulting in highly variable postoperative glucose control. No other study has yet investigated the effect of preoperative carbohydrate loading on glucose control the first days after the bariatric surgery in patients who have poor glycemic control

DETAILED DESCRIPTION:
Bariatric surgery allows weight loss and obesity related comorbidities remission. In patients with type 2 diabetes (T2D), glucose intolerance (GI) and metabolic syndrome (MS), weight loss surgery improves glucose control more than medications and/or life style intervention. This approach is gaining acceptance even in patients with mild obesity and indications are now rapidly growing. Roux en Y gastric bypass (RYGB) and Sleeve Gastrectomy (SG) the gold standard operations for treating T2D, lower glycemia often very rapidly and sometime profoundly. The responsible mechanisms are not completely understood and guidelines for the early management of T2D and GI following bariatric surgery are lacking, resulting in highly variable postoperative glucose control.

The recent use of a pre-operative carbohydrate loading compared to fasting has been shown to improve the early recovery after surgical procedures by reducing the profound stress response following surgery and allowing a better postoperative blood glucose regulation by lowering insulin resistance.

Metabolic stress and insulin resistance follow major surgery. The resulting post-operative hyperglycaemia is associated with increased morbidity as well as mortality. In non-diabetic patients, avoiding pre-operative fastening substantially reduces post-operative stress and insulin resistance. A pre-operative carbohydrate load improves post-operative glycaemic control, most likely by inducing endogenous insulin release before the onset of surgery. This sets the metabolic state of the patient in a fed rather than a fasted state at the time of surgery. Metabolic reactions to surgical stress are thereby markedly reduced not only resulting in a reduced risk for hyperglycaemia during post-operative nutrition but also retained lean body mass, improved muscle strength and nitrogen economy.

The oral preparation used is a carbohydrate-rich clear beverage containing mainly polymers of carbohydrates to minimize the osmotic load. The drink, in addition to its metabolic effect, improves patient well-being (thirst, hunger, anxiety) pre-operatively. Oral preload is considered the first element in the surgical pathway to reduce patients' stress with the aim of early return to oral diet, mobility and recovery as soon as possible after surgery and had a significant effect on reducing complications and improving wellbeing.

Patients with GI and T2D are at particular risk of impaired glycaemic control peri-operatively. Most of the studies using pre-operative carbohydrate loading were performed on non-diabetic patients. A considerable number of patients going through bariatric surgery suffer from GI or T2D (respectively 30% and 15% in our experience), this patient group has been denied initially for the pre-operative carbohydrate drink because of fear of slow gastric emptying and impaired glycaemic control. We are aware of only one study that evaluated the suitability for diabetic patients to have preload drinks pre-operatively . Gustafsson et al explored the possibility of providing pre-operative carbohydrate loading in patients with mild T2D without neuropathy or delayed gastric emptying (as autonomic neuropathy is a likely cause of delayed gastric function in diabetes). In this study, T2D patients (n=25) showed no signs of hyperglycaemia. However, the wider spectrum of diabetic patients was not evaluated. Can et al. also evaluated the effects of pre-operative pre-loading in patients with or without insulin resistance. This differed from other studies, which had previously excluded those with known insulin resistance. This study included 34 cholecystectomy or thyroidectomy patients showed that the temporal pattern of plasma glucose in patients with insulin resistance who were given preload drinks pre-operatively was similar to that of patients without insulin resistance. These studies suggest that there might be a benefit without risk of hyperglycaemia to give to type-2 diabetic (and GI) patients a preload along with their usual diabetic medication. No other study has yet investigated the effect of preoperative carbohydrate loading on glucose control the first days after the bariatric surgery in patients who have poor glycemic control. Furthermore, most bariatric surgery studies include only late postoperative evaluations of glucose control, such as those made after 7 days or more.

The main hypothesis of this study is that pre-operative carbohydrate loading compared to fasting will optimize the overall pattern of postoperative glucose profile evidenced by Continuous Glucose Monitoring (CGM) with a greater impact in the first few days after surgery on lowering mean glycaemia and glycemic variability in patients with glucose intolerance.

The primary aim is to evaluate the mean of all blood glucose measures of CGM over 24-h period after surgery in patients receiving pre-operative carbohydrate loading in comparison with standard 6h fasting. The mean of all glucose measures over 24- h of CGM (around 288) reflects overall glucose control including fasting and postprandial state. It have been chose to study this early period to minimize any confounding effects of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery planned (RYGB or SG)
* BMI at least 35 kg/m2 with comorbidity that can be improved after surgery(including cardiovascular disease including high blood pressure, obstructive sleep apnea syndrome and other severe respiratory disorders, severe metabolic disorders, particularly type 2 diabetes, disabling osteoarticular disease, steatohepatitis non-alcoholic)
* Glucose Intolerance as defined by the American Diabetes Association (ADA Diabetes Care 2017)
* Negative pregnancy test
* Informed consent
* Patient with social insurance

Exclusion Criteria:

* Patients receiving insulin therapy
* Previous bariatric surgery
* Definite symptoms of gastroparesis assessed by Gastroparesis Cardinal Symptoms Index (GCSI)*. Values of score ≥ 1.90 will be chosen as definite symptoms of gastroparesis.
* Pregnant or breastfeeding woman, persons deprived of their liberty, persons under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mean blood glucose level of CGM over 24-h period beginning the day after surgery in patients receiving pre-operative carbohydrate loading in comparison with standard 6h fasting | Day 1 after surgery
  mean blood glucose level over 24h at D1 after surgery, as assessed by CGM

SECONDARY OUTCOMES:
mean blood glucose value | preoperative, Day2 and Day 3 after surgery, Day 4 to 6 after surgery, 3 months after surgery
  mean blood glucose level over 24h, as assessed by CGM, during preoperative period, day2 and day 3 after surgery, day4 to 6 after surgery and at 3 months
post prandial peak glucose (Gmax) | preoperative, Day1 after surgery, Day2 and Day 3 after surgery, Day 4 to 6 after surgery, 3 months after surgery
  post prandial peak glucose (Gmax) will be assessed by CGM over 24h period, during preoperative period, day2 and day 3 after surgery, day4 to 6 after surgery and at 3 months
the time spent in hyperglycemic range (> 12 mmol / L) | preoperative, Day1 after surgery, Day2 and Day 3 after surgery, Day 4 to 6 after surgery, 3 months after surgery
  the time spent in hyperglycemic range will be assessed by CGM over 24h period, during preoperative period, day2 and day 3 after surgery, day4 to 6 after surgery and at 3 months
time spent in hypoglycemic range (<2.4 mmol / L) | preoperative, Day1 after surgery, Day2 and Day 3 after surgery, Day 4 to 6 after surgery, 3 months after surgery
  the time spent in hypoglycemic range (<2.4 mmol / L)will be assessed by CGM over 24h period, during preoperative period, day2 and day 3 after surgery, day4 to 6 after surgery and at 3 months
total area under the glucose curve (AUC20) | preoperative, Day1 after surgery, Day2 and Day 3 after surgery, Day 4 to 6 after surgery, 3 months after surgery
  total area under the glucose curve (AUC20) will be calculated using CGM data over 24h period, during preoperative period, day2 and day 3 after surgery, day4 to 6 after surgery and at 3 months
glycemic instability as measured by standard deviation of differences in values of glucose separated by a number of hours (between 1 and 24 hours) (Continuous overall net glycemic action: CONGA). | preoperative, Day1 after surgery, Day2 and Day 3 after surgery, Day 4 to 6 after surgery, 3 months after surgery
  glycemic instability as measured by standard deviation of differences in values of glucose separated by a number of hours (between 1 and 24 hours) (Continuous overall net glycemic action: CONGA) will be calculated using CGM data over 24h period, during preoperative period, day2 and day 3 after surgery, day4 to 6 after surgery and at 3 months
Rate of patients wit blood glucose levels within a target range (120 to 180 mg / dL [6.67 to 10 mmol / L]) during the perioperative period | preoperative, Day1 after surgery, Day2 and Day 3 after surgery, Day 4 to 6 after surgery, 3 months after surgery
  rate of patients with blood glucose level within a larger range on CGM values
Length of hospital stays after surgery | at 1 month after surgery
  regarding the initial bariatric procedure
Rate of early surgical perioperative complications | at 1 month after surgery
  within the 30 days after surgery
Rate of patients needing antibiotic therapy | at 1 month after surgery
  within the 30 days after surgery
Rate of patients needing reoperation | at 1 month after surgery
  within the 30 days after surgery
Rate of patients normoglycemic at 3 months, defined as blood glucose below 5.5mMol/L and HbA1c of less than 6% in the absence of any antidiabetic medication | at 3 months after surgery
  rate of normoglycemic patients

CONTACTS AND LOCATIONS:
Overall Officials: Robert Caiazzo, MD,PhD, Principal Investigator — University Hospital, Lille